CLINICAL TRIAL: NCT01673061
Title: Vapocoolant Spray as a Novel Local Anesthetic for Cutaneous Abscess Incision and Drainage
Brief Title: Vapocoolant Spray for Numbing Small Boils Before Incision and Drainage
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Vapocoolant not effective controlling pain compared with Lidocaine.
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN 4405
Record Dates: First submitted 2012-08-14; First posted 2012-08-27 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2014-06

CONDITIONS: Abscess
Keywords: Abscess; Boils; Anesthetics, Local; Lidocaine; Vapocoolant; 1,1,1,3,3-Pentafluoropropane; 1,1,1,2-Tetrafluoroethane
MeSH Terms: conditions — Abscess; Furunculosis | interventions — Lidocaine; Epinephrine; 1,1,1,3,3-pentafluoropropane; norflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine injection will be used for anesthesia prior to incision and drainage. 2% Lidocaine with epinephrine will be injected into the abscess site. Amount injected will be per physician discretion.
  Interventions: Drug: Lidocaine
- Vapocoolant (Active Comparator): Vapocoolant spray will be used for anesthesia prior to incision and drainage. The spray will be administered to the abscess site for a duration of 2 seconds, from a distance of 12 cm.
  Interventions: Drug: Vapocoolant

INTERVENTIONS:
Drug: Lidocaine — See associated Arm Description
  Other Names: Lidocaine with Epinephrine
  Arms: Lidocaine
Drug: Vapocoolant — See associated Arm Description
  Other Names: Gebauer's Pain Ease; Numbing Spray; 1,1,1,3,3-Pentafluoropropane; 1,1,1,2-Tetrafluoroethane
  Arms: Vapocoolant

SUMMARY:
Cutaneous abscesses (boils) are collections of pus or infection in the skin, and are a frequent reason for emergency department visits. The only proven cure for abscesses is cutting them open and allowing the infection to drain, but this procedure is often painful. Currently, the usual method of pain control is to inject a numbing medication (lidocaine) into the site, but this injection itself is often painful and sometimes does not offer full pain relief. Although there has been some research into the use of non-injected numbing agents as another option, no studies have looked at the use of numbing sprays (vapocoolant) in this context specifically. The hypothesis of this study is that numbing spray is as good as injected numbing medication at relieving pain in patients having small abscesses opened and drained. This theory will be tested by taking two groups of patients having small abscesses drained in the Emergency Department, and assigning one group to get a numbing injection, and the other to get a numbing spray. Their levels of pain and satisfaction will be recorded before, during, and after the procedure, and the two groups will be compared.

DETAILED DESCRIPTION:
Hypotheses: Patients would have a similar amount of pain with incision and drainage using local infiltration of anesthetic as with application of a vapocoolant spray and the pain of the administration of anesthesia would be similar or reduced with the use of the vapocoolant spray.

Specific aims: 1.Non-inferiority in pain of anesthesia administration and incision and drainage of small abscesses by finding no significant difference of patient pain as measured on the VRNS scale.

2. Show that patients were willing to undergo anesthesia again with a vapocoolant spray as assesed by the Likert scale Long term goals- To implement the use of vapocoolant sprays as an alternative form of anesthesia for incision and drainage of abscesses

The primary outcome measure for this study would be the finding of no significant difference in the pain as measured by the VRNS between the two arms for administration of anesthesia. Secondary measures would be finding no significant difference in VRNS for incisional and drainage, and change in VRNS from presentation to anesthesia, and to incision and drainage, willingness of the patient to choose the allocated sprayin the future, and unexpected events.

Initial medical assessment will be made by an attending/senior resident in accordance with established clinical procedures, including the history, physical examination, and vital signs. If by clinical assessment the patients meet eligibility criteria, then they will be approached by a research associate for screening, informed consent process, enrollment in the study, and data collection. Following the screening questionnaire, the research associate will hold thorough discussion about the study. The patients will be given as much time as they require to understand and make an informed decision. A formal written consent will be obtained if patients agree to participate. After the patient understands and signs the informed consent form, they will be randomized to either the placebo group or treatment group by using a randomization scheme. The treating physician will measure erythema and induration using a measuring tape, estimate the amount of fluctuance as small, moderate, or large, and note the location of the abscess. Once randomized, subjects will be given a VRNS scale to rate their pain upon initial presentation The treating physician will clean the abscess with chlorhexidine solution then either spray the skin overlying the abscess with 1,1,1,3,3-Pentafluoropropane and 1,1,1,2-Tetrafluoroethane spray (Gebauer's Pain Ease® Medium Stream Spray) at a distance of 12 cm from the site for a duration of 2 seconds or infiltrate the abscess with 2% lidocaine with epinepherine (amount determinted by treating physician). Any reactions to the vapocoolant administration will be noted. The abscess will then be incised with a No. 11 surgical scalpel, and a cotton tipped applicator will be used to break up loculations within the abscess cavity. The method of I&D, and decision to probe to break-up loculations will be standardized, but the degree of probing, and decision to pack will be left to the discretion of the treating physician. Subjects will be asked by the research assistant to describe the discomfort of the abscess using the Visual Numerical Rating Scale (VRNS) during vapocoolant administration, during incision of the abscess, and after the procedure is complete.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old
* Able to consent
* Has cutaneous abscess less than or equal to 2 centimeters requiring incision and drainage in the Emergency Department

Exclusion Criteria:

* Less than 18 years old
* Unable to consent
* Pregnant or breastfeeding
* Prisoner or in police custody
* Known sensitivity to vapocoolant or lidocaine
* Cold hypersensitivity
* Chronic steroid use
* Peripheral neuropathy
* Diabetes
* HIV
* Malignancy
* Immunosuppressive state
* Sickle cell disease
* Sarcoidosis
* Abscess greater than 2 centimeters in any dimension
* Abscess requiring procedural sedation and analgesia for incision and drainage, or further intervention outside the Emergency Department
* Abscess located on the hands, feet, face, or perineal areas
* Pilonidal cyst
* hidradenitis suppurativa
* Not a good candidate per attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D'Orazio, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer AJ, Richman PB, Kowalska A, Thode HC Jr. Comparison of patient and practitioner assessments of pain from commonly performed emergency department procedures. Ann Emerg Med. 1999 Jun;33(6):652-8. PMID 10339680
- [Background] Hijazi R, Taylor D, Richardson J. Effect of topical alkane vapocoolant spray on pain with intravenous cannulation in patients in emergency departments: randomised double blind placebo controlled trial. BMJ. 2009 Feb 10;338:b215. doi: 10.1136/bmj.b215. PMID 19208703
- [Background] Costello M, Ramundo M, Christopher NC, Powell KR. Ethyl vinyl chloride vapocoolant spray fails to decrease pain associated with intravenous cannulation in children. Clin Pediatr (Phila). 2006 Sep;45(7):628-32. doi: 10.1177/0009922806291013. PMID 16928840
- [Background] Cohen Reis E, Holubkov R. Vapocoolant spray is equally effective as EMLA cream in reducing immunization pain in school-aged children. Pediatrics. 1997 Dec;100(6):E5. doi: 10.1542/peds.100.6.e5. PMID 9374583
- [Background] Mawhorter S, Daugherty L, Ford A, Hughes R, Metzger D, Easley K. Topical vapocoolant quickly and effectively reduces vaccine-associated pain: results of a randomized, single-blinded, placebo-controlled study. J Travel Med. 2004 Sep-Oct;11(5):267-72. doi: 10.2310/7060.2004.19101. PMID 15544709
- [Background] Cannon CR, Replogle B. Fine-needle aspiration biopsy: is anesthesia necessary? Otolaryngol Head Neck Surg. 1999 Apr;120(4):458-9. PMID 10187933
- [Background] Browne J, Awad I, Plant R, McAdoo J, Shorten G. Topical amethocaine (Ametop) is superior to EMLA for intravenous cannulation. Eutectic mixture of local anesthetics. Can J Anaesth. 1999 Nov;46(11):1014-8. doi: 10.1007/BF03013194. PMID 10566919
- [Background] Biro P, Meier T, Cummins AS. Comparison of topical anaesthesia methods for venous cannulation in adults. Eur J Pain. 1997;1(1):37-42. doi: 10.1016/s1090-3801(97)90051-3. PMID 15102427
- [Background] Rosier EM, Iadarola MJ, Coghill RC. Reproducibility of pain measurement and pain perception. Pain. 2002 Jul;98(1-2):205-16. doi: 10.1016/s0304-3959(02)00048-9. PMID 12098633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Pre-assignment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Period: Overall Study
Arm/Group | Lidocaine | Vapocoolant
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Vapocoolant | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: VNRS Pain Scale - Anesthetic Administration
Description: Visual Numeric Rating Scale (VNRS) for pain level at time of anesthetic administration on Day 1.
Time Frame: Once, on Day 1, at time of anesthetic administration
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: VNRS Pain Scale - Incision and Drainage
Description: Visual Numeric Rating Scale (VNRS) for pain level during incision and drainage of the abscess on Day 1.
Time Frame: Once, on Day 1, at time of incision and drainage
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in VNRS - From Pre-anesthesia to Administration of Anesthesia
Description: Difference between the VNRS pain scale values collected just prior to anesthesia administration, and at the moment of anesthesia administration, on Day 1.
Time Frame: Once, on Day 1
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in VNRS - From Pre-anesthesia to Post-procedure
Description: Difference between the VNRS pain scale values collected just prior to anesthesia administration, and at after all aspects of incision and drainage are complete, on Day 1.
Time Frame: Once, on Day 1
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Willingness to Use Method of Anesthesia in the Future
Description: Willingness of the subject to use their assigned method of anesthesia again if they were to require the same procedure in the future. Measured once on Day 1.
Time Frame: Once, on Day 1
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Unexpected Events
Description: Any unexpected events that would occur during study period, including adverse events, on Day 1.
Time Frame: Measured continuosly from consent to discharge, on Day 1.
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0
Description: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | Lidocaine | Vapocoolant
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes